CLINICAL TRIAL: NCT06382766
Title: Skeletal Muscle Ultrasonography in Detection of Malnutrition and Prediction of The Outcome Among Critically Ill Children Attending Assiut University Children Hospital
Brief Title: Skeletal Muscle Ultrasonography in Detection of Malnutrition
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Hussin Mohamed, assisstant lecturer of pediatrics, Assiut University
Other Study IDs: SMU in malnutrition
Record Dates: First submitted 2024-02-18; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Skeletal Muscle Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Skeletal Muscle Ultrasonography — Skeletal Muscle Ultrasonography in Detection of Malnutrition and Prediction of The Outcome among critically ill children

SUMMARY:
* To detect the role of Skeletal Muscle Ultrasonography in Detection of Malnutrition and Prediction of The Outcome among critically ill children.
* To assess the accuracy and validity of muscle ultrasonography in assessment of the nutritional status of critically ill child compared with other different nutritional assessment tools .

DETAILED DESCRIPTION:
Under nutrition is a public health problem worldwide, particularly among children under-five. Globally in 2020, about 149.2 million (22% of children under-five) and 45.4 million (6.7% of children under-five) were estimated to be stunted and wasted respectively . Undernutrition equally accounts for about 3.1 million deaths (45% of all deaths) among children under-five annually . This burden, however, is disproportionately borne by the African continent. In effect, two out of five (41% or 61.4 million children) stunted children and more than a quarter (27% or 12.1 million children) of all wasted children under-five live in the African continent. This burden varied across the country, greatest in rural localities and areas with ongoing humanitarian crisis.

Pediatric intensive care unit (PICU) admission rates for undernutrition in critically sick children range from 8.1 to 71.7%, despite variations in nutritional indices, the presence of chronic illness, age, and critical illness severity . Critically ill children can become undernourished more quickly than adults due to their lower body fat and muscle mass and higher per kilogram resting energy requirements. Complications from undernutrition can include more frequent infections, longer length of stay (LOS), and morbidity.

Underweight children admitted to the pediatric intensive care unit (PICU) have a higher mortality and PICU LOS, which increase with increasing severity of underweight. In light of this, early detection of undernutrition and the observation of nutritional status degradation might result in fast and appropriate nutritional therapies, which may improve clinical outcomes. Additionally, because most critically ill patients have reduced nutritional reserves, iatrogenic underfeeding and increasing malnutrition are further encouraged by prolonged fasting and frequent feeding pauses during intensive care unit (ICU) and hospital stays No single objective marker can be used to reliably predict protein-energy malnutrition or risk of nutrition-related complications in children; an assessment encompassing several markers is necessary. The diagnosis of malnutrition can be based on 6 different domains: (1) insufficient food and nutrition intake compared with nutrition requirements, (2) weight loss over time, (3) loss of muscle mass, (4) loss of fat mass, (5) fluid accumulation, and (6) measurably diminished grip strength. Hence, no single measure (either anthropometric or laboratory) by itself is an ideal measure of malnutrition.

Anthropometric measurements are essential components of nutrition screening and assessment of pediatric patients. The use of proper equipment, accurate measurement techniques, and appropriate reference data are necessary for obtaining and interpreting anthropometric data. Accurate height and length measurements can be difficult to obtain in ambulatory children and in some clinical situations (such as trauma, burn, and surgical patients who require the use of traction, castings, or dressings for large body wounds), accurate anthropometric measurements such as weight and height may be more difficult or impossible to obtain. Preliminary evidence suggests that muscle wasting also occurs in critically ill children, which could affect intensive care unit (ICU) course or long-term growth and development in children.

Identification of muscle wasting would thus be important in critically ill children, so as to be able to appropriately target optimal nutrition and physical interventions to reduce muscle wasting and risk of poor outcomes in these high-risk children. However, identifying muscle changes can be challenging in clinical practice. Current methods available, such as mid-arm circumference, may not accurately reflect muscle changes, while other methods such as computerized tomography (CT) or magnetic resonance imaging (MRI) are not easily conducted at bedside. Recently, ultrasonography has been used in adult critical care to visualize abnormalities and changes in muscle throughout the course of the ICU stay. Ultrasonography, an imaging technique that uses reflections of high-frequency sound waves directed at tissues, is noninvasive, fast, and cost-effective, and it has been suggested as a possible nutrition assessment tool in critically ill patients. Muscle ultrasound enables early detection of skeletal muscle wasting, which is associated with histological changes in muscle as well as functional impairment in adults. Muscle ultrasonography has also traditionally been used to quantify and qualify muscle morphology in pediatric populations, especially children with neuromuscular diseases.

A necessary first step is identification of the most appropriate muscle group. A variety of body sites have been studied in children, the most common of which include the quadriceps, gastrocnemius, tibia, biceps, and forearm.

Muscles are studied either individually (eg, rectus femoris) or in combination with others (eg, rectus femoris and vastus intermedius) in single or various limbs.

Using a variety of muscle groups allowed for a more comprehensive assessment of whole-body nutrition assessment of children, which required ultrasound measurement of both fat and muscle layer thickness (MLT) at 9 sites, including anterior and posterior upper and lower limbs, as well as subscapular and abdominal areas. Equations using these measurements produced fat and muscle mass estimations comparable to that measured using more sophisticated imaging methods such as MRI and dual-energy x-ray absorptiometry (DXA). However, as whole-body ultrasound measurements may require a significant amount of time, some longitudinal studies have used single limbs for ultrasound measurements. In children with cancer in whom reduced lean body mass could negatively affect disease outcomes, monthly ultrasound demonstrated changes in quadriceps thickness throughout the course of cancer therapy. This suggests that, unlike in the diagnosis of neuromuscular disease, a single muscle group may be sufficient to monitor changes in body composition over time in certain groups of pediatric patients.

Both upper and lower body muscle wasting has been reported in critically ill children,and some adult data suggest that muscle wasting affects lower limbs more than upper limbs.

The quadriceps alone has also been used to monitor muscle changes in critically ill adults. Measurements of the thickness of the rectus femoris, vastus intermedius, and vastus lateralis and cross-sectional area (CSA) of the rectus femoris on alternate days demonstrate an overall decreasing trend in the first 10 days of critical illness.The quadriceps is the most commonly studied lower limb muscle in children.

Loss of muscle mass is associated with poor clinical outcomes. Patients who develop muscle wasting have higher risk of intensive care unit (ICU) acquired weakness , increased length of ICU stay and loss of muscle mass during the frst week of ICU stay is associated with increased mortality risk . Weakness and fatigue are persisting symptoms which have a negative impact on the quality of life of critical illness survivors.

Thus muscle ultrasound may add benefit in early detection of undernutrition in practice ,so this study will be conducted to explore the accuracy of muscle ultrasound in detection of undernutrition in PICU in comparison to the traditional nutritional assessment tools and to explore its impact on prognosis of such cases.

ELIGIBILITY:
Inclusion Criteria:

* Acute critically ill infants and children aged > 1month- 5 years .

Exclusion Criteria:

* Neonates less than 1 month .
* Children with muscle disorders .
* Children with multiple congenital anomlies, genetic or chromosomal diseases.
* Children with chronic illness or comorbid condition (T.B, diabetes, malignancy, etc..) .
* children missed for follow up.

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Acute critically ill infants and children aged > 1month- 5 years attending Assiut University Children Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
accuracy of Skeletal Muscle Ultrasonography in Detection of Malnutrition and Prediction of The Outcome among critically ill children comared with other traditional nutritional assessment tools . | one year
  skeletal muscle ultrasonography every 3 days.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garcia GH, Fu MC, Dines DM, Craig EV, Gulotta LV. Malnutrition: a marker for increased complications, mortality, and length of stay after total shoulder arthroplasty. J Shoulder Elbow Surg. 2016 Feb;25(2):193-200. doi: 10.1016/j.jse.2015.07.034. Epub 2015 Oct 9. PMID 26456427
- [Result] Mehta NM, Duggan CP. Nutritional deficiencies during critical illness. Pediatr Clin North Am. 2009 Oct;56(5):1143-60. doi: 10.1016/j.pcl.2009.06.007. PMID 19931068
- [Result] Abera EG, Sime H. The prevalence of malnutrition among critically ill children: a systematic review and meta-analysis. BMC Pediatr. 2023 Nov 21;23(1):583. doi: 10.1186/s12887-023-04419-x. PMID 37986053
- [Result] Kasaye HK, Bobo FT, Yilma MT, Woldie M. Poor nutrition for under-five children from poor households in Ethiopia: Evidence from 2016 Demographic and Health Survey. PLoS One. 2019 Dec 20;14(12):e0225996. doi: 10.1371/journal.pone.0225996. eCollection 2019. PMID 31860689
- [Result] Ngassa AB, Meriki HD, Mbanga CM, Nzefa LD, Mbhenyane X, Tambe AB. Key predictors of undernutrition among children 6-59 months in the Buea Health District of the Southwest region of Cameroon: a cross sectional community-based survey. BMC Nutr. 2022 Dec 13;8(1):148. doi: 10.1186/s40795-022-00646-0. PMID 36514089